CLINICAL TRIAL: NCT05180760
Title: Effectiveness of a Smartphone App in Promoting Weight Loss in Patients With Non-alcoholic Fatty Liver Disease: a Pilot Multi-centre Randomized Controlled Trial
Brief Title: Smartphone App for Non-alcoholic Fatty Liver Disease
Acronym: AppLiver
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HKU01
Record Dates: First submitted 2021-12-01; First posted 2022-01-06 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: non-alcoholic fatty liver disease; telemedicine; mobile health; self-management
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone app arm (Active Comparator): Use the dedicated smartphone app for NAFLD patients
  Interventions: Behavioral: Smartphone app use
- Standard of care (Other): Standard of care
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Smartphone app use — Smartphone app use in the active arm
  Arms: Smartphone app arm
Behavioral: Standard of care — Standard of care
  Arms: Standard of care

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a disease spectrum that encompasses excessive liver deposition of fat (NAFL), non-alcoholic steatohepatitis (NASH), and NASH cirrhosis. NAFLD is regarded as the hepatic manifestation of metabolic syndrome and is currently the most common etiology for chronic liver disease worldwide, affecting 25% of the adult population globally. It is estimated that cirrhosis and liver-related death occur in 20% and 12%, respectively, over a 10-year period in patients with NAFLD. The incidence of decompensated cirrhosis and hepatocellular carcinoma (HCC) due to NAFLD are increasing with time. In United States, the number of patient listing for liver transplantation (LT) due to NAFLD has surpassed that of from chronic viral hepatitis and is currently the second leading cause for LT waitlist overall. Locally, the prevalence of NAFLD is estimated to be 42% according to a health census in healthy blood donors in Hong Kong, and up to 13.5% healthy subjects will develop new onset NAFLD in 3-5 years of follow-up.

Clearly, NAFLD is a chronic liver disease with alarmingly high prevalence that warrants attention. Despite the high prevalence and potential to develop serious liver-related morbidity, there are currently no approved drugs for patients with NAFLD. To achieve resolution of steatohepatitis and improvement of liver fibrosis, weight loss appears to be the only effective means.

This study is aimed to evaluate the effectiveness of a self-developed smartphone app for achieving weight loss in Chinese adults with non-alcoholic fatty-liver disease (NAFLD) at 12 months. Endorsed by the WHO, mobile technology is being increasingly used to promote health. There is a lack of research on the use of mobile technology for promoting weight loss in Chinese NAFLD patients.

DETAILED DESCRIPTION:
The Investigators formed a multi-disciplinary team consisting of hepatologist, computer scientist, dietitian and endocrinologist. The investigators hypothesize that NAFLD subjects who use the dedicated smartphone app will achieve more weight loss than subjects who are managed with standard of care (SOC) without smartphone app.

The present study is a multi-center, two-arm randomized, placebo-controlled, 1:1 trial to examine the effectiveness of a self-developed simple-to-use smartphone app for NAFLD patients. The smartphone app consists of elements that track health data, provide health education, estimate calorie intake and energy expenditure. Anthropometric measurements, blood tests, transient elastography, and bioelectrical impedance analysis will be performed at baseline and 12 months. The intervention is either Smartphone app vs SOC. The main outcome measures will include changes in body weight, liver fat, liver enzyme, muscle mass, lipid and glucose profile.

ELIGIBILITY:
Inclusion Criteria:

* known NAFLD
* able to read and understand Chinese
* owns a compatible smartphone
* without major cognitive impairment.

Exclusion Criteria:

* on SGLT-2 inhibitors, GLP-1 agonists, or thiazolidinediones
* patients with cirrhosis
* patients who are pregnant
* patients on special diet or with special dietary requirement (e.g. vegan, gluten free)
* patients with heavy alcohol use (≥20 grams/ day for women or ≥30 grams/ day for men)
* history of HCC or LT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | 12 months
  Body weight of the participants will be measured at baseline and 12 months

SECONDARY OUTCOMES:
Reduction in hepatic steatosis | 12 months
  Hepatic steatosis will be quantified by transient elastography as expressed by controlled attenuation parameter (CAP)
ALT normalization | 12 months
  ALT as part of liver biochemistry will be measured at baseline and 12 months
Reversal of sarcopenia | 12 months
  Skeletal muscle mass will be quantified by bioelectrical analysis. Sarcopenia is common among subjects with NAFLD and is defined according to international guidelines.
Changes in lipid profile | 12 months
  Fasting lipid profile will be measured at baseline and 12 months
Changes in glucose levels | 12 months
  Fasting glucose levels will be measured at baseline and 12 months
Visceral fat reduction | 12 months
  Visceral fat will be assessed using bioelectrical analysis machine at baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Yi Mak, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Select A State Or Province, China

IPD SHARING:
Plan to Share IPD: No